CLINICAL TRIAL: NCT01768754
Title: Repeatability and Utility of the Usual and Fast Walking Speeds in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Walking Speeds in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Roger Goldstein, Director, Respiratory Medicine, West Park Healthcare Centre
Other Study IDs: Goldstein_Walk_COPD
Record Dates: First submitted 2013-01-09; First posted 2013-01-15 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Exercise testing; Functional status; Pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD patients: Usual and Fast Walking Speeds
  Interventions: Behavioral: Usual and Fast Walking Speeds

INTERVENTIONS:
Behavioral: Usual and Fast Walking Speeds — Stable patients with chronic obstructive pulmonary disease will demonstrate their usual and fast walking speeds over a 30 m course, with speed calculated over the middle 10 m using optical sensors. The test will be repeated after a 5 minute rest; this procedure will then be repeated on two subsequent days, at the same time of day, within one week.

SUMMARY:
A growing body of evidence suggests that in individuals with chronic lung disease their walk speed is related to their daily function and quality of life. It is possible to assess their usual (routine) and fast walking speeds by getting them to walk in a flat hallway.

In individuals with chronic lung disease, we anticipate that their usual walk speed will be helpful in exercise prescription and use in multidimensional scoring systems. However, it is important to first determine the measurement properties of these two walk speeds.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and spirometric diagnosis of COPD
* Able to provide written informed consent

Exclusion Criteria:

* Unstable cardiovascular disease
* Acute respiratory exacerbation within 4 weeks
* Neurologic or orthopedic limitation to walking
* Inability to comprehend instructions in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable moderate-severe COPD will be recruited from those under the care of a respirologist at West Park Health Care Centre
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Coefficient of repeatability for usual and fast walk speeds | At baseline and over 1 week period.
  Participants will be asked to demonstrate their usual and fast walk speeds over the middle 10 meters of a 30 meter straight track using optical sensors and a hand-held stopwatch. Participants will be instructed to walk at their 'usual' and 'fast' speeds as standardized instructions. The walk test will be repeated after a 5 minute rest and then repeated on two subsequent days, at the same time of day, within one week. This will be simply observational in nature with no planned intervention aside for controlling walking environment.
  The primary outcome is going to report a change in walk speeds from baseline and at 1 and 2 days using repeated measures as described by Bland and Altman (reference below).

SECONDARY OUTCOMES:
Agreement in walk speeds between optical sensors and stopwatch | Baseline and over 1 week of testing.
  Assess agreement between the use of optical sensors and stop watch time for the usual and fast walk speeds.
Agreement in the Bode Index using six minute walk distance and usual walk speed. | Baseline
  To assess agreement in the calculated Bode Index using the six minute walk distance versus estimated usual walk speed distance over 6 minutes.

OTHER OUTCOMES:
Precision of achieving a targeted endurance time using the usual and fast walking speeds. | Baseline
  The usual and fast walk speeds will be used to predict the test speed for a high-intensity constant-speed endurance test that will achieve an acceptable endurance time of 2-15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Goldstein, MD, FRCPC, Principal Investigator — Westpark Healthcare Centre
Locations (1):
- Westpark Health Care Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Bland JM, Altman DG. Measuring agreement in method comparison studies. Stat Methods Med Res. 1999 Jun;8(2):135-60. doi: 10.1177/096228029900800204. PMID 10501650